CLINICAL TRIAL: NCT04768556
Title: Assessment of Brain Activity Associated With Inhibition of Action in Attention-deficit Hyperactivity Disorder
Brief Title: Brain Activity Associated With Inhibition of Action in Attention-deficit
Acronym: INHIB'MOV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/20/0252
Record Dates: First submitted 2021-02-05; First posted 2021-02-24 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Attention Deficit; Hyperactivity Disorder
Keywords: KEYWORDS: Inhibitory control; time-frequency
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: This study is pathophysiological, monocentric, comparative, and controlled with 3 groups compared: ADHD patients, control patients (negative diagnosis of ADHD), and healthy volunteers.
  The three groups will complete the same protocol, in the same manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ADHD group (Experimental): ADHD group: 20 participants having received a positive diagnosis of ADHD
  Interventions: Other: EEG experimental sessions 1; Other: EEG experimental sessions 2
- Control group 1 (Other): Control group 1: 20 participants having received a negative diagnosis of ADHD
  Interventions: Other: EEG experimental sessions 1; Other: EEG experimental sessions 2
- Control group 2 (Other): Control group 2: 20 participants as healthy volunteers
  Interventions: Other: EEG experimental sessions 1; Other: EEG experimental sessions 2

INTERVENTIONS:
Other: EEG experimental sessions 1 — An EEG experimentation session on the stop-signal task of inhibiting a prepared discrete graphic action.
Other: EEG experimental sessions 2 — An EEG experimentation session on the stop-signal task of inhibiting an ongoing rhythmic action

SUMMARY:
Inhibitory control allows individuals to suppress unwanted actions and to resist irrelevant stimuli. It is thought to be a core deficit in Attention-deficit/hyperactivity disorder (ADHD). The present study aims at evaluating this deficit in adults with ADHD. Executive and inhibitory capacities, as well as the neural mechanisms underlying inhibitory control, will be assessed in adults with ADHD and two control groups of participants.

DETAILED DESCRIPTION:
ADHD is a psychiatric disorder characterized by symptoms of inattention, hyperactivity, and impulsivity (DSM-V, 2013). An impairment of inhibitory control has been suggested as the primary deficit in children with ADHD, which is thought to cause secondary impairments in executive functioning. A few studies investigated executive capacities in adults with ADHD. Specifically, an impairment in action inhibition has been reported in ADHD participants. Moreover, inhibition of action is often associated with distinctive electroencephalographic (EEG) correlates. The present study aim at combining both novel inhibitory control measurement techniques and EEG analysis in temporal and frequency domains to assess the sensitivity and the specificity of an inhibitory deficit in adults with ADHD. This is part of an improvement in the procedures for diagnosing ADHD syndrome and its functional evaluation.

The study will analyze the EEG activity associated with two stop-signal tasks requiring inhibitory capacities. A set of other cognitive skills will also be evaluated during a neuropsychological assessment. The results of ADHD patients will be compared with those of a control group (healthy volunteers) to assess the sensitivity of an inhibition deficit to the disorder. These same results will also be compared with those of a second control group (patients with a negative diagnosis of ADHD) to assess the specificity of the inhibitory deficit.

This experimental strategy results in the involvement of three groups of participants (ADHD patients and two control groups) in three visits (neuropsychological assessment and two EEG sessions).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50,

  * Visual, auditory (authorized apparatus), motor skills suitable for the proper realization of neuropsychological tests,
  * Being right-handed,
  * Free, informed and written consent signed by the participant and the investigator
  * Person affiliated or beneficiary of a social security scheme.
* For the ADHD group:

  * Diagnosis of ADHD according to DSM-V criteria (APA, 2013),

For the patient control group:

• Patient who consulted for a cognitive complaint and for whom the diagnosis of ADHD was rejected according to the criteria of DSM-V (APA, 2013).

Exclusion Criteria:

* General or progressive neurological disease resulting in cognitive impairment (multiple sclerosis, Parkinson's disease, stroke, etc.),
* Insufficient linguistic level in French to participate in neuropsychological assessment,
* Patient placed under judicial protection or under another protective regime,
* Severe depression according to DSM-V criteria (APA, 2013),
* Autism spectrum disorder, developmental coordination disorder.

  -For the healthy voluntary control group:
* Presence of a cognitive complaint or pathology which may impair his cognitive functions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
EEG correlates of inhibition | 2 weeks
  The main objective of this study is to evaluate, by electrophysiological measures, the presence of a deficit of action inhibition in adults with ADHD. To this end, the EEG correlates of inhibition will be compared between participants in the three groups. Thus, the ERP (N2 / P3) and ERSP (Theta, Delta) variations observed in terms of amplitude and latency in the stop-signal task tests will be computed in each of the three groups.

SECONDARY OUTCOMES:
Inhibition performance from a rhythmic-action task | 2 weeks
  The inhibition performance from a rhythmic-action task, expressed as stop-signal reaction time (SSRT, in ms). This latency is measured by identifying a statistical deviation evoked by the STOP signal in the participants' movement on a graphic tablet (following the procedure described in Hervault et al., 2019).
Inhibition performance from a discrete-action task | 2 weeks
  The inhibition performance from a discrete-action task, expressed as an SSRT (in ms). According to the horse-race model of inhibition, this latency is estimated based on the response time and the response probability obtained by the participants when responding to the GO and STOP stimuli used in the task (following recent guidelines from Verbruggen et al., 2019).

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie PARIENTE, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Toulouse Purpan University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No